CLINICAL TRIAL: NCT07331324
Title: The Coma Family Program (COMA-F): A Multi-site Clinical Trial of a Resilience Program for Caregivers of Patients With Severe Acute Brain Injury
Brief Title: The Coma Family Program (COMA-F): A Resilience Program for Caregivers of Patients With Severe Acute Brain Injury
Acronym: COMA-F
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alexander Presciutti, Member of the Faculty, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P003235
Record Dates: First submitted 2025-12-16; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Caregiver Distress; Emotional Distress; Caregivers; Resilience; Coma; Brain Injury
Keywords: caregivers; emotional distress; caregiver burden; resilience; coma; severe acute brain injury; mindfulness
MeSH Terms: conditions — Coma; Brain Injuries; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coma Family Program 1 (Experimental): This arm provides skills training to manage distress, uncertainty, and long-term caregiving challenges.
  Interventions: Behavioral: Coma Family Program 1
- Coma Family Program 2 (Placebo Comparator): This arm involves providing education about managing caregiving distress, uncertainty, and long-term challenges.
  Interventions: Behavioral: Coma Family Program 2

INTERVENTIONS:
Behavioral: Coma Family Program 1 — This intervention provides skills training to manage distress, uncertainty, and long-term caregiving challenges.
  Arms: Coma Family Program 1
Behavioral: Coma Family Program 2 — This involves education (but no skills training) about managing caregiving distress, uncertainty, and long-term challenges.
  Arms: Coma Family Program 2

SUMMARY:
The purpose of this research study is to see if two different psychosocial programs for caregivers of patients with severe acute brain injuries are able to improve caregiver mental health.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older - study population
2. English fluency and literacy - measures and intervention are in English
3. Screens positive for emotional distress on either depression or anxiety subscales (>7) of the Hospital Anxiety and Depression scale - study population (caregivers must be at-risk for chronic distress via heightened acute distress)
4. Confirmed by the clinical team as the primary caregiver of a patient who has been admitted to an intensive care unit (ICU) with a severe acute brain injury with the following characteristics:

   1. 18 years or older - study population
   2. Admitted with ischemic stroke, intracerebral hemorrhage, subarachnoid hemorrhage, traumatic brain injury, or hypoxic-ischemic encephalopathy - study population
   3. Glasgow Coma Scale score below 9 (in judgement of the clinical team) while not intubated or an inability to follow meaningful commands while intubated at any point during the hospitalization for > 24 consecutive hours due to the brain injury itself and not a confounding factor (e.g., sedation or seizures) - study population
   4. Still alive in ICU at the time the clinical team approaches the caregiver about possible recruitment - excludes caregivers of those that passed away as would require a different intervention (e.g., grieving intervention)
   5. Has been committed to or has already received long-term life-sustaining treatments including tracheostomy and/or percutaneous endoscopic or surgical gastrostomy tube placement (trach or PEG) - study population; at time of enrollment patients can be in various early stages of cognitive/functional recovery from initial coma, but all were severe enough to require trach and/or PEG
   6. Has a prognosis for survival of greater than 3 months and does not have a concurrent diagnosis of a terminal illness or injury as judged by the clinical team - as in "d"; such caregivers would require different intervention
   7. Is still in ICU or has been transferred to a lower level of care (e.g., stepdown) for <7 days at the time of consent - study population; we aim to begin the intervention when caregivers are acutely distressed in the context of the patient's ICU stay or shortly after the ICU stay (i.e., within 7 days of leaving)

Exclusion Criteria:

* 1. Serious mental illness, substance misuse, or active suicidal intent or plan - requires higher level of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Hospital anxiety and depression scale | baseline, 6-weeks, and 3-month follow-up
  Measures anxiety and depression. Anxiety and depression sub scales each range from 0 (minimum) to 21 (maximum) with higher scores meaning worse outcome.

SECONDARY OUTCOMES:
Posttraumatic stress disorder checklist-5 | baseline, 6-weeks, and 3-month follow-up
  measures posttraumatic stress symptoms. Scores range from 0 (minimum) to 80 (maximum) with higher scores indicating worse outcome.
World Health Organization Quality of Life-Short Form | baseline, 6-weeks, and 3-month follow-up
  Measures quality of life across four domains, physical, psychological, social, and environmental. Scores on each sub scale range from 0 (minimum) to 100 (maximum) with higher scores indicating better outcome.

OTHER OUTCOMES:
Cognitive and Affective Mindfulness Scale | baseline, 6-weeks, and 3-month follow-up
  measures dispositional mindfulness. Scores range from 12 (minimum) to 48 (maximum), with higher scores indicating better outcome (greater dispositional mindfulness).
Applied Mindfulness Process Scale | baseline, 6-weeks, and 3-month follow-up
  measures applied mindfulness. Scores range from 0 (minimum) to 60 (maximum) with higher scores indicating better outcome (more frequent application of mindfulness skills in daily life).
Measure of Current Status-A | baseline, 6-weeks, and 3-month follow-up
  measures adaptive coping. Scores range from 0 (minimum) to 4 (maximum) with higher scores indicating better outcome (better use of adaptive coping skills).
Intolerance of Uncertainty Scale Short Form | baseline, 6-weeks, and 3-month follow-up
  Measures intolerance of uncertainty. Scores range from 12 (minimum) to 60 (maximum) with higher scores indicating worse outcome (greater intolerance of uncertainty).
Zarit Burden Interview Short Form | baseline, 6-weeks, and 3-month follow-up
  Measures caregiver burden. Scores range from 0 (minimum) to 48 (maximum) with higher scores indicating worse outcome (greater caregiver burden).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Data includes caregiver demographic characteristics, health characteristics (quality of life), and outcome assessments (e.g., emotional distress, coping, mindfulness, etc). These measures will be self-reported. We will also collect limited quantitative data extracted from patients' medical charts (diagnosis, age, race, ethnicity). All data will be de-identified and preserved for at least seven years after closing the study with IRB. Quantitative datasets will be made available via the Vivli database.
Supporting Information: Study Protocol, ICF
Time Frame: All de-identified data will be preserved for at least seven years after closing the study with IRB.
Access Criteria: The de-identified quantitative dataset will be made freely available for requests that are ethically sound.